CLINICAL TRIAL: NCT06991530
Title: Effect of Low Molecular Weight Heparin in Freeze-thaw Embryo Transfer Cycles in Women With Recurrent Implantation Failure
Status: Completed | Type: Observational
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Linlin Cui, professor, The Second Hospital of Shandong University
Other Study IDs: KYLL2025342
Record Dates: First submitted 2025-04-29; First posted 2025-05-28 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Low Molecular Weight Heparin; Recurrent Implantation Failure; FET; IVF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LMWH group: the LMWH group received injections of 4100 IU/d LMWH from the day of transplant
  Interventions: Drug: Low Molecular Weight Heparine
- Control group: the control group received the routine luteal support protocol (without LMWH use)

INTERVENTIONS:
Drug: Low Molecular Weight Heparine — the LMWH group received injections of 4100 IU/d LMWH from the day of transplant
  Groups: LMWH group

SUMMARY:
Recurrent implantation failure (RIF) is considered a tough problem in assisted reproductive technology (ART) without effective treatments. The effect of low molecular weight heparin (LMWH) in pregnancy outcomes is controversial. In addition, there are few reports on the role of LMWH in population with RIF performing freeze-thaw embryo transfer (FET) cycles. The purpose of this study is to evaluate the effect of LMWH on pregnancy outcomes in women with FET cycles.

ELIGIBILITY:
Inclusion Criteria:

* Women under or equal to the age of 40 when oocytes were retrieved;
* The history of at least 2 failed fresh embryo transfer/FET cycles and cumulative transfer of ≥ 3 high-quality embryos or cumulative transfer of ≥ 2 blastocysts;
* Planning to FET after IVF or ICSI cycles

Exclusion Criteria:

* Women with untreated hydrosalpinx, uterine cavity occupying lesions (uterine adhesions, submucous fibroids, endometrial polyps, et al.);
* Women with abnormal anatomical structure of uterus (unicornuate uterus, bipedal uterus, et al.);
* Women with endometrial thickness (EMT) < 6mm on the day of transplantation;
* Women or their partner with abnormal chromosome karyotype (not including chromosome polymorphisms);
* Women with the history of recurrent spontaneous abortion (RSA);
* Women with a history of autoimmune or coagulation disorders;
* Women with contraindications to LMWH

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study analyzed the data from the hospital electronic database for patients undergoing FET between January, 2021 and November, 2024, a total of 392 transplant cycles, who undergoing at least two IVF or ICSI cycles from the Second Hospital of Shandong University.
Sampling Method: Non-Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | from transplantation to delivery (assessed up to 40 weeks of gestation)
  The number of ongoing pregnancies divided by the number of women who received a transfer

SECONDARY OUTCOMES:
biochemical pregnancy rate | from transplantation to delivery (assessed up to 40 weeks of gestation)
  The number of biochemical pregnancy cycles divided by the number of transplantation cycles
clinical pregnancy rate | from transplantation to delivery (assessed up to 40 weeks of gestation)
  The number of clinical pregnancies divided by the number of women who received a transfer
ectopic pregnancy rate | from transplantation to delivery (assessed up to 40 weeks of gestation)
  The number of ectopic pregnancies divided by the number of women who received a transfer
Miscarriage rate | from transplantation to delivery (assessed up to 40 weeks of gestation)
  The number of miscarriages divided by the number of clinical pregnancies

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
The investigators fully acknowledge the significance of data sharing as stipulated by SCI journals. However, owing to the policies and confidentiality agreements adhered to in our laboratory, the investigators regretfully cannot furnish the raw data. Nevertheless, the investigators have meticulously presented a comprehensive account of the experimental design, analysis, results, and the procedures employed for data analysis and processing.